CLINICAL TRIAL: NCT07101510
Title: Effectiveness of Video-assisted Cardiopulmonary Resuscitation Under Special Circumstances: a Randomized Controlled Simulation Study
Brief Title: V-CPR Under Special Circumstances
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pecs (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: V-CPR special circumstances
Record Dates: First submitted 2025-07-28; First posted 2025-08-03 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-07

CONDITIONS: Cardiac Arrest (CA)
Keywords: cardiac arrest; video-assisted CPR; cardiopulmonary resuscitation; V-CPR; special circumstances; dispatcher
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants will be informed about their group assignment post-randomization but will be blinded to the study's aims. The dispatcher and the simulation operator will be briefed on their specific tasks but will remain blinded to the study hypotheses and outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- sV-CPR (Experimental): Participants perform video-assisted CPR based on the European Resuscitation Council (ERC) 2021 guidelines.
  Interventions: Behavioral: sV-CPR
- V-CPR (Active Comparator): Participants perform video-assisted CPR based on the European Resuscitation Council (ERC) 2021 guidelines.
  Interventions: Behavioral: V-CPR
- T-CPR (Active Comparator): Participants perform telephone-assisted CPR based on the European Resuscitation Council (ERC) 2021 guidelines.
  Interventions: Behavioral: T-CPR
- sT-CPR (Experimental): Participants perform telephone-assisted CPR based on the European Resuscitation Council (ERC) 2021 guidelines.
  Interventions: Behavioral: sT-CPR

INTERVENTIONS:
Behavioral: sV-CPR — In the sV-CPR group, participants manage a simulated cardiac arrest scenario alone. They perform CPR while establishing a video connection with a dispatcher located in another room using a smartphone. To simulate challenging conditions, they must carry out the task in near-total darkness, with the phone's flashlight as the only light source.
  Arms: sV-CPR
Behavioral: V-CPR — In the V-CPR group, participants manage a simulated cardiac arrest scenario alone. They perform CPR while establishing a video connection with a dispatcher located in another room using a smartphone.
  Arms: V-CPR
Behavioral: T-CPR — In the T-CPR group, participants manage a simulated cardiac arrest scenario alone. They perform CPR while establishing a telephone connection with a dispatcher located in another room using a smartphone (vocal communication only).
  Arms: T-CPR
Behavioral: sT-CPR — In the sT-CPR group, participants manage a simulated cardiac arrest scenario alone. They perform CPR while establishing a telephone connection with a dispatcher located in another room using a smartphone (vocal communication only). To simulate challenging conditions, they must carry out the task in higher environmental noises (traffic), generated by a loudspeaker.
  Arms: sT-CPR

SUMMARY:
Out-of-hospital cardiac arrest (OHCA) remains a major cause of death globally, with bystander CPR rates varying widely (13-82%) despite public health efforts. Early recognition, EMS activation, and immediate CPR are key to survival, often beginning with a layperson guided by an emergency dispatcher.

Telephone-assisted CPR (T-CPR), where dispatchers give verbal instructions, is common but limited-dispatchers can't see the scene or correct CPR technique. In contrast, video-assisted CPR (V-CPR) enables visual feedback, potentially improving performance in areas like compression rate and hand placement. However, evidence is mixed regarding its effect on compression depth, and initiating a video call may introduce delays.

While V-CPR's technical benefits have been studied, little is known about how real-world distractions-like noise or poor lighting-affect its effectiveness. Our simulation study aimed to compare T-CPR and V-CPR under both ideal and challenging conditions to assess the impact of environmental factors on layperson CPR quality and dispatcher support.

DETAILED DESCRIPTION:
Out-of-hospital cardiac arrest (OHCA) remains a major global health concern and one of the leading causes of mortality in industrialized nations. Despite various public health initiatives aimed at increasing layperson engagement in early intervention, bystander cardiopulmonary resuscitation (CPR) rates continue to vary widely across countries, ranging from 13% to 82%. Survival after OHCA is strongly associated with the early recognition of cardiac arrest, rapid activation of emergency medical services (EMS), and immediate initiation of effective CPR. In most cases, the first responder is a layperson who contacts the emergency dispatcher-making dispatcher-assisted CPR a critical link in the chain of survival.

Telephone-assisted CPR (T-CPR), where the dispatcher provides audio instructions, is a widely adopted and effective method to initiate life-saving efforts. However, the lack of visual feedback limits its potential: the dispatcher cannot observe the victim's condition, the responder's technique, or the scene dynamics. As a result, certain errors may go uncorrected, and the quality of CPR may be suboptimal.

With advancements in communication technology, real-time video communication between dispatchers and callers has become feasible. Video-assisted CPR (V-CPR) allows dispatchers to visually assess the situation, provide tailored feedback, and correct lay responder errors during the intervention. Several simulation studies have demonstrated that V-CPR can improve CPR performance compared to T-CPR, particularly in terms of compression rate, hand placement, and technique. However, the evidence regarding its superiority in achieving guideline-recommended compression depth remains mixed. Furthermore, the added complexity of initiating a video call and ensuring optimal camera positioning can delay CPR initiation and affect its effectiveness.

While prior studies have explored the technical feasibility and clinical benefits of V-CPR, the influence of environmental and situational variables-such as background noise, poor lighting conditions, or the presence of distractions-remains underexplored. These factors are highly relevant in real-world emergencies and may impact both the lay responder's performance and the dispatcher's ability to guide the process effectively.

Our study aimed to address this gap by conducting a simulation trial to compare the effectiveness of T-CPR and V-CPR under both ideal and environmentally challenging conditions. By systematically examining the impact of common distracting factors, our goal was to better understand the limitations and potential of video-assisted emergency guidance in realistic layperson resuscitation scenarios.

ELIGIBILITY:
Inclusion Criteria:

* healthy voluntear

Exclusion Criteria:

* healthcare professionals (paramedics, nurses, etc.)
* pregnant women
* people with cardio-pulmonary and musculoskeletal diseases or any other impairment that would risk harm for the volunteer while performing CPR for 2 minutes
* physical and/or psychological disabilities
* technical issue during data collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2025-08-10 (Actual); Primary Completion 2025-09-10 (Actual); Study Completion 2025-09-10 (Actual)

PRIMARY OUTCOMES:
Chest compression depth | During procedure.
  Chest compression depth will be evaluated by a manikin connected to a CPR software.

SECONDARY OUTCOMES:
Chest compression rate | During procedure
  Chest compression rate will be evaluated by a manikin connected to a CPR software.
Hand position during chest compression. | During procedure
  Hand position during chest compression will be evaluated by observation.

OTHER OUTCOMES:
Attitude of participants | Immediately after the CPR procedure (within 15 minutes)
  Subjective feelings after performing CPR based on a short survey using Likert-scale based queries (lower numbers indicate worse, higher score indicates better opinion).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pécs, Pécs, Hungary